CLINICAL TRIAL: NCT04432311
Title: A Randomized Controlled Trial Comparing a Group-based Guided Self-help Approach to Pure Self-help for the Treatment of Binge Eating Disorder
Brief Title: Comparing a Group-based Guided Self-help Approach to Pure Self-help for the Treatment of BED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Aaron Keshen, Psychiatrist, Principal Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFT 2.0
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Binge Eating Disorder
Keywords: Binge Eating Disorder; Binge Focused Therapy (BFT); Self-Help; Guided Self-Help
MeSH Terms: conditions — Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binge Focused Therapy (BFT) (Experimental): Guided self-help - Three online group sessions, homework, and self-guided check-ins to monitor continued progress and/or signs of relapse.
  Interventions: Behavioral: Binge Focused Therapy (BFT)
- CBT Unguided Self Help (CBT USH) (Active Comparator): Pure self-help - The use of the book Overcoming Binge Eating and its associated homework.
  Interventions: Behavioral: CBT Unguided Self Help (CBT USH)

INTERVENTIONS:
Behavioral: Binge Focused Therapy (BFT) — The BFT group will be provided Binge Focused Therapy, a group-based, guided-self help intervention. Participants in this group will attend three online group sessions spread over six weeks (Week 1, Week 2, and Week 6) and complete homework between sessions. Following Session 3, there is a four week period where participants complete self-guided check-ins once per week to monitor continued progress and/or signs of relapse.
  Arms: Binge Focused Therapy (BFT)
Behavioral: CBT Unguided Self Help (CBT USH) — The CBT USH group will be provided with the book, Overcoming Binge Eating by C. Fairburn, which is a well-established self-help book used to help individuals understand binge eating and control binge eating behaviours. After participants receive the book, they will have 10 weeks to read it and work through the exercises provided in the book.
  Arms: CBT Unguided Self Help (CBT USH)

SUMMARY:
Binge eating disorder (BED) is the most common eating disorder in adults, affecting 2.8% of the population. The disorder is characterized by recurrent episodes of binge eating which are not followed by inappropriate compensatory behaviours such as self-induced vomiting. BED is associated with an increased risk of health complications, significant impairment to social and occupational functioning, and reduced quality of life. Despite the negative consequences associated with this disorder, standard therapy for BED is often inaccessible and costly.

To address the limitations of standard therapy for BED our research team has developed Binge Focused Therapy (BFT) as an innovative, guided self-help approach to BED treatment. BFT was derived from elements of "The Brain Over Binge Recovery Guide" by Kathryn Hansen, which incorporates fundamental aspects of Acceptance and Commitment Therapy, Dialectical Behaviour Therapy, Motivational Enhancement Therapy, and addictions treatment. We further streamlined this approach into a protocol that can be delivered by non eating disorder specialists (e.g., honours psychology students, nurses, occupational therapists).

In 2018, our research team conducted a proof-of-concept pilot study with a sample of 40 individuals with BED. Unpublished results of this uncontrolled study indicated that the sample experienced significant reductions in binge episodes per month, binge eating severity, general eating disorder symptomology, and improved confidence in changing binge eating behaviours.

Although the results from this small, uncontrolled, proof-of-concept study are encouraging, qualitative and quantitative data highlighted several aspects of the BFT intervention that could be altered and tested in a randomized controlled trial that compares BFT to an active comparator.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for Diagnostic and Statistical Manual of Mental Disorders (5th Edition) diagnosis of BED (mild-extreme) as per Eating Disorder Examination - Mild severity will be modified from a minimum of 1 objective binge episode/week to 2 objective binge episodes per week
* Age 18 or older
* Access to computer with internet connection and webcam that can be used in a private area
* Virtually signed informed consent form

Exclusion Criteria:

* Currently receiving psychotherapy/treatment for BED (as determined by PI)
* Self-reported Body Mass Index on pre-screening questionnaire < 20 kg/m2
* Dose change of a psychotropic medication used for the treatment of BED (e.g., Vyvanse, topiramate, antidepressants) or any medication that could have an effect on appetite/binging (e.g., Saxenda) within 4 weeks of study inclusion (as determined by PI)
* Insufficient knowledge of English
* Previously participated in proof-of-concept BFT study
* Previously read Overcoming Binge Eating by C. Fairburn and implemented strategies presented in the book (as determined by PI)
* Serious physical illness (e.g., severe uncontrolled insulin dependent diabetes) (as determined by PI)
* Currently pregnant
* Scores greater than 20 on the Quick Inventory of Depressive Symptomatology Self-Report and PI determines participant is significantly depressed (as determined by PI)
* Currently experiencing serious issues with alcohol or drugs (as determined by PI)
* Currently engaging in self-harm behaviours (as determined by PI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Binge Eating Symptomology | Baseline to Post-Treatment (10 week)
  This will be measured using the global score generated from the Binge Eating Scale (BES). The BES is a 16-item measure, each item has 3-4 coded responses. The total score ranges from 0-46, where a higher score indicates greater binge eating severity.

SECONDARY OUTCOMES:
Binge Eating Symptomology | 6 week, 6-month follow-up, 12-month follow-up
  This will be measured using the global score generated from the Binge Eating Scale (BES). The BES is a 16-item measure, each item has 3-4 coded responses. The total score ranges from 0-46, where a higher score indicates greater binge eating severity.
Binge Eating Frequency | Baseline, 6 week, 10 week, 6-month follow-up, 12-month follow-up
  Self reported changes in Binge Eating Frequency over past 28 days will be measured using Item 15 from the Eating Disorder Examination Questionnaire 6.0 (EDE-Q; Fairburn & Beglin, 1994) which inquires about the number of days with objective binge episodes over the past 28 days.
Eating Disorder Symptomology (Eating Disorder Examination Questionnaire) | Baseline, 6 week, 10 week, 6-month follow-up, 12-month follow-up
  Self reported changes in Eating Disorder Symptomology will be measured using the global score generated from the EDE-Q (Fairburn & Beglin, 1994). The EDE-Q is a 28-item measure that assesses four areas of eating disorder psychopathology (eating concern, shape concern, weight concern, dietary restraint). Each item uses a Likert scale ranging from 0 (lowest frequency/severity) to 6 (highest frequency/severity). The global score ranges from 0-6 where higher scores indicate greater impairment. The global score is obtained using the mean of the four subscales.
Clinical Impairment | Baseline, 6 week, 10 week, 6-month follow-up, 12-month follow-up
  Self reported changes in clinical impairment will be measured using the Clinical Impairment Assessment Questionnaire (CIA; Bohn & Fairburn, 2008). This is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features over the past 28 days. Each item is ranked on a 0-3 scale (0 being "not at all" and 3 being "a lot"). Total scores range from 0-48, with higher scores indicating greater clinical impairment.
Confidence to Change Binge Eating | Baseline, 6 week, 10 week, 6-month follow-up, 12-month follow-up
  Confidence to Change Binge Eating will be measured using the question, "On a scale from 1 to 10, how confident are you that you can change your binge eating if you wanted to?", with higher scores indicating greater confidence. This question assesses perceived confidence in ability to change binge eating.
Abstinence | Week 10, 6-month follow-up, 12-month follow-up
  Abstinence is defined as a 100% reduction in binge episodes in the 28 days prior to collecting outcome measures.
Remission | Week 10, 6-month follow-up, 12-month follow-up
  Remission is defined as meeting criteria for abstinence (100% reduction in binge episodes in the 28 days prior to collecting outcome measures) in addition to having EDEQ global score less than or equal to 2.77 (Fairburn & Beglin, 1994).
Intervention Adherence | Week 6, Week 10
  Intervention adherence for participants in the BFT group will be based on session attendance. Completers will be defined as anyone who completes Session 1 and at least one other session. Adherence questionnaires at Week 6 and Week 10 time points inquire about which aspects of the intervention outside of the sessions have been used.
  Intervention adherence for participants in the CBT USH group will be calculated using questionnaires provided at both the Week 6 and Week 10 time points that inquire about which chapters have been read and which "CBT Steps" have been completed thus far. Completers will be defined as anyone who indicates that they have read Chapters 1, 4, 5, and 'Getting Ready', and completed Step 1 through Step 3.
Participant Expectations | Pre-Intervention, Week 1
  This will be measured using the Credibility and Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000). The CEQ is a six item self-report measure that measures treatment expectancy and rationale credibility of therapeutic interventions. Each item is scored on a 1-9 Likert-type scale or as a percentage rating from 0% to 100% in increments of 10%. Higher scores indicate greater credibility/expectancy of the intervention.
Satisfaction with Intervention | Week 10
  Participants in both groups will respond to developed Likert-style and open-ended questions asking about their perceptions of their assigned program. Each Likert item is ranked on a scale from 1-9. Higher total scores indicate greater satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Keshen, MD, FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Heath Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No